CLINICAL TRIAL: NCT00644904
Title: A Phase I/II Dose-Escalation Trial of Vitamin D3 With Calcium Supplementation in Patients With Multiple Sclerosis
Brief Title: Safety Trial of High Dose Oral Vitamin D3 With Calcium in Multiple Sclerosis
Acronym: VitD4MS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Direct MS-Proactive Charity (Unknown); Multiple Sclerosis Society of Canada (Other)
Responsible Party: Dr. Paul O'Connor, St. Michael's Hospital, Division of Neurology, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB05-147
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Vitamin D; Safety
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Starting dose of 4,000 IU per day of Vitamin D3 titrating up to a dose of 40,000 IU per day of Vitamin D3 by month six. In the second six-month part of the trial, patients titrate back down to 4,000 IU per day of Vitamin D3 and then discontinue it completely at the end of the 12 month trial period.
  Interventions: Dietary Supplement: Vitamin D3
- Control (Other): Patients are allowed to supplement with up to 4,000 IU per day of Vitamin D3 if desired.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3
  Arms: Treatment
Dietary Supplement: Vitamin D3
  Arms: Control

SUMMARY:
Vitamin D likely plays a role in the geography of Multiple Sclerosis (MS), and patients at risk and with MS have relatively low Vitamin D levels compared to their normal counterparts.

This trial examines the safety of high dose oral Vitamin D3 titrated up to a maximum of 40,000 IU per day over a 12 month period. Fifty patients matched for MS and non-MS characteristics will be divided into two groups: one group receiving the high dose Vitamin D regimen, and the other restricted to a maximum of 4000 IU per day. The hypothesis is that patients with MS can tolerate seemingly high doses of Vitamin D3 without adverse events and/or calcium-related abnormalities. It is also hypothesized that those receiving the higher doses will demonstrate improved relapse and disability status compared to controls, and that the treatment group will show improved markers of bone health and immune indicators of reduced inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite MS
* Age 18-55
* EDSS 0-6.5

Exclusion Criteria:

* EDSS => 7.0
* Current Vitamin D3 use >4000 IU/d
* Baseline (25(OH)D) level <20 mmol/L (frank deficiency) and >150 mmol/L
* Pregnancy or inability/unwillingness to use contraception
* History of cardiac arrhythmia
* History of renal disease and nephrolithiasis
* History of granulomatous disease or lymphoma
* Relapse activity or steroid use in the past 60 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2006-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Serum calcium | at each dose change

SECONDARY OUTCOMES:
Serum 25(OH)D | at each dose change
EDSS | at screening vs. end of trial
N-telopeptide (bone marker)
ALP/AST/ALT | at each dose change
Creatinine/urea | at each dose change
EKG | at screening and end of trial
Renal ultrasound | at screening, mid-trial and end of trial
Cytokine profile/MMP/lymphocyte response assay
Annualized relapse rate | year prior to trial versus year of trial
PTH | at each dose change

CONTACTS AND LOCATIONS:
Overall Officials: Jodie M Burton, MD, Principal Investigator — St. Michael's Hospital, University of Toronto; Paul W O'Connor, MD, MSc, Principal Investigator — St. Michael's Hospital, University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Kimball SM, Ursell MR, O'Connor P, Vieth R. Safety of vitamin D3 in adults with multiple sclerosis. Am J Clin Nutr. 2007 Sep;86(3):645-51. doi: 10.1093/ajcn/86.3.645. PMID 17823429
- [Derived] Kimball S, Vieth R, Dosch HM, Bar-Or A, Cheung R, Gagne D, O'Connor P, D'Souza C, Ursell M, Burton JM. Cholecalciferol plus calcium suppresses abnormal PBMC reactivity in patients with multiple sclerosis. J Clin Endocrinol Metab. 2011 Sep;96(9):2826-34. doi: 10.1210/jc.2011-0325. Epub 2011 Jun 22. PMID 21697250
- [Derived] Kimball SM, Burton JM, O'Connor PG, Vieth R. Urinary calcium response to high dose vitamin D3 with calcium supplementation in patients with multiple sclerosis. Clin Biochem. 2011 Jul;44(10-11):930-2. doi: 10.1016/j.clinbiochem.2011.04.017. Epub 2011 May 5. PMID 21570386